CLINICAL TRIAL: NCT04380792
Title: Prevalence of DVT or PE in Patients Infected With COVID-19 Admitted to Hospital (SCREENING Study)
Brief Title: Prevalence of DVT or PE in Patients Infected With COVID-19 Admitted to Hospital
Acronym: SCREENING
Status: Completed | Type: Observational
Sponsor: Manuel Monreal (Other)
Responsible Party: Sponsor-Investigator, Manuel Monreal, Professor of Internal Medicine, Foundation for the study of VTE diseases. (FUENTE)
Organization: Foundation for the study of VTE diseases. (FUENTE) (Other)
Other Study IDs: SCREENING042020
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objectives are:

* To establish the prevalence of deep venous thrombosis through ultrasonography in Patients infected with COVID-19 admitted to hospital.
* To identify patients with higher risk of deep venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with COVID-19.
* Admission to hospital.

Exclusion Criteria:

* Patients treated with ECMO (Extracorporeal membrane oxygenation).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients infected with COVID-19 admitted to hospital
Sampling Method: Non-Probability Sample
Enrollment: 2497 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
VTE events and complications | 30 days
  Study endpoints are clinically recognized (and objectively confirmed) recurrences of VTE, major and minor bleeding complications, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Monreal, Study Chair — Germans Trias i Pujol Hospital
Locations (1):
- Manuel Monreal, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided